CLINICAL TRIAL: NCT04576728
Title: A Randomized, Placebo-controlled, Double-blind, Multi-center, Phase II Trial Investigating the Efficacy and Safety of Trimodulin (BT588) as add-on Therapy to Standard of Care in Adult Subjects With Severe COVID-19
Brief Title: Efficacy and Safety of Trimodulin in Subjects With Severe COVID-19
Acronym: ESsCOVID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biotest (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 998
Record Dates: First submitted 2020-09-24; First posted 2020-10-06 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Covid19
Keywords: Covid19; Severe community acquired pneumonia; Acute Respiratory Distress Syndrome; SARS-CoV-2; Severe Corona Virus Disease
MeSH Terms: conditions — COVID-19; Community-Acquired Pneumonia; Respiratory Distress Syndrome | interventions — trimodulin

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized on a 1:1 basis either to trimodulin or to placebo treatment stratified by center.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All bottles will be indistinguishable.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trimodulin (Experimental): Trimodulin (human IgM, IgA, IgG solution) for intravenous (IV) administration.
  Interventions: Drug: Trimodulin
- Placebo (Placebo Comparator): Human albumin 1%
  Interventions: Other: Placebo (human albumin 1%)

INTERVENTIONS:
Drug: Trimodulin — IMP will be administered via IV infusion on 5 consecutive days.
  Other Names: BT588
  Arms: Trimodulin
Other: Placebo (human albumin 1%) — IMP will be administered via IV infusion on 5 consecutive days.
  Arms: Placebo

SUMMARY:
The objectives of the trial are to evaluate the efficacy and safety of trimodulin as add-on therapy to standard of care (SoC) compared to placebo treatment in adult hospitalized subjects with severe COVID-19.

Additionally, pharmacodynamic (PD) and pharmacokinetic (PK) properties of trimodulin will be evaluated in all subjects.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind, multi-center, phase II trial investigating the efficacy and safety of trimodulin compared to placebo treatment, as add-on therapy to SoC in adult subjects with severe COVID-19. Severe COVID-19 patients with need for non-invasive ventilation or high flow oxygen and with dysregulated inflammatory responses demonstrated by an elevated CRP level, will be enrolled.

Subjects will be randomized to receive either trimodulin or placebo on a 1:1 basis, stratified by center. Investigational Medicinal Product (IMP) treatments will be blinded. Subjects will be administered IMP once daily on five consecutive days (day 1 through day 5) as add-on therapy to SoC. The subsequent follow-up phase comprises 23 [+3] days (day 6 through day 28) followed by an end-of-trial visit/ telephone call on day 29 [+3]. For evaluation of this trial, a 9-category ordinal scale will be used. The primary aim of trimodulin treatment in the enrolled severely ill patients with a score of 5, is to prevent their clinical deterioration to a critical disease stage (score 6-7, e.g. requiring invasive mechanical ventilation or ECMO) and death (score 8). Accordingly, a composite primary efficacy endpoint reflecting the deterioration / mortality rate is used.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the subject or legally authorized representative or informed verbal or administration consent due to pandemic situation, in compliance with all local legal requirements.
2. Male or female subject ≥18 years of age.
3. Laboratory-confirmed SARS-CoV-2 infection from a test done in a respiratory tract sample within the last 5 days at screening.
4. Diagnosis of community-acquired severe COVID-19 within 10 days after hospital-admission, with severe defined as:

   Need for non-invasive ventilation (NIV), or high-flow oxygen therapy (score =5 on the 9-category ordinal scale).

   At least one of the following clinical respiratory parameters is fulfilled: dyspnea, respiratory frequency ≥30/min, SpO2 ≤93%, 100 mmHg < PaO2/FiO2 ≤300 mmHg, and/or lung infiltrates >50% within 24 to 48 hours.

   At least one measurement of C-reactive protein ≥50 mg/L within 36 hours prior to start of treatment.
5. Subject must receive SoC treatment for COVID-19.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Subjects that deteriorated to score >5 on the 9-category ordinal scale (e.g. receiving invasive mechanical ventilation (IMV), and/or extracorporeal membrane oxygenation (ECMO)) or subjects that improved to score <5 prior to randomization.
3. Severe neutropenia (neutrophil count <500/mm³) assessed within 24 hours prior to start of treatment.
4. Thrombocytopenia (platelet count <30,000/mm³) assessed within 24 hours prior to start of treatment.
5. Hemoglobin <7g/dL assessed within 24 hours prior to start of treatment.
6. Known hemolysis.
7. Known thrombosis or thromboembolic events (TEEs) or known medical history of TEEs (e.g. cerebrovascular accidents, transient ischemic attack, myocardial infarction, pulmonary embolism, and deep vein thrombosis) within the previous 3 months or those subjects particularly at risk for TEEs (e.g. history of thrombophilia, permanent immobilization, or permanent paralysis of the lower extremities) caused by other reasons than COVID-19.
8. Subject on dialysis or with severe renal impairment, estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m² assessed within 24 hours prior to start of treatment (details in Appendix 3: Estimated Glomerular Filtration Rate).
9. Subject with end stage renal disease (ESRD), or known primary focal segmental glomerulosclerosis (FSGS).
10. Known severe lung diseases interfering with COVID-19 therapy (e.g. severe interstitial lung disease, cystic fibrosis, idiopathic pulmonary fibrosis, active tuberculosis, chronically infected bronchiectasis, or active lung cancer).
11. Known decompensated heart failure (New York Heart Association class III-IV).
12. Known pre-existing hepatic cirrhosis, severe hepatic impairment (Child Pugh C score ≥9 points), or hepatocellular carcinoma.
13. Known intolerance to proteins of human origin or known allergic reactions to components of trimodulin.
14. Selective, absolute immunoglobulin A (IgA) deficiency with known antibodies to IgA.
15. Known treatment for thorax/head/neck/hematologic malignancies in the last 12 months.
16. Known human immunodeficiency virus infection.
17. Life expectancy of less than 90 days, according to the Investigator's clinical judgment, because of medical conditions neither related to COVID-19 nor to associated medical complications.
18. Obesity (body mass index ≥40 kg/m²), a body weight of more than 123 kg, or anorexia (body mass index <16 kg/m²).
19. Known immunosuppressive treatment other than acute treatment for COVID-19 (e.g. transplant recipient, subject with autoimmune disease).
20. Known treatment with polyvalent immunoglobulin preparations, any type of blood product, or any type of interferon during the last 21 days before entering the trial.
21. Participation in another interventional clinical trial within 30 days before entering, or during the trial, or previous participation in this clinical trial.
22. Employee or direct relative of an employee of the contract research organization, the trial site, or Biotest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
Clinical detoriation rate | Between day 6 and day 29
  Percentage of subjects with a change of clinical status to score 6 or 7 on the 9-category ordinal scale
28-day all-cause mortality rate | Between day 1 and day 29
  Percentage of subjects with a change to score 8 on the 9-category ordinal scale

SECONDARY OUTCOMES:
Clinical deterioration rate | Days 1-29 and days 6-29
  Percentage of subjects with a change to score 6-7
28-days all-cause mortality rate on day 29 | Day 29
  Percentage of subjects with score=8, assessed at the end-of-trial visit on day 29 [+3].
Time to clinical deterioration | Time Frame: between Days 1-29 and days 6-29
  Number of days to first change from score 5 (enrollment) to score 6-7
Time to Mortality | Time Frame: between Day 1 and day 29
  Number of days to change to score =8
Proportion of subjects in each of the 9-categories of the ordinal scale | Days 7, 14, 21, 29
  Number of patients by score on specific study days
Time to clinical improvement | Day 29
  Number of days to change to score 4 (mild disease, with supplemental oxygen) or score 3 (mild disease, no supplemental oxygen)
Proportion of subjects with score ≤2 | Day 29
  Proporation of subjects that improved to score ≤2
Days on IMV | Until day 29
  Number of calendar days on IMV until day 29
Days without oxygen supply | Until day 29
  Number of calendar days without any form of oxygen support until day 29
Time to discontinuation from any form of oxygen supply | Until day 29
  Time to definite stop of any form of additional oxygenation, irrespective of short interruptions
Proportion of subjects without any form of oxygen supply | Day 29
  Proportion of subjects that improved to not requiring supplemental oxygen.
Hospital-free-days | Until day 29
  Calendar days between hospital discharge and day 29
SARS-CoV-2 status | Until day 29
  Time to SARS-CoV-2 negative status
Adverse events (AEs), treatment-emergent AEs (TEAEs), AEs of special interest, infusional TEAEs | Until day 29
  Number, severity, causality, outcome, and seriousness of all. AE, TEAEs that led to permanent withdrawal of IMP, and TEAEs that led to discontinuation of the trial.
TEAEs | Until day 29
  Number of all infusion related TEAEs
SAEs | Until day 29
  Number, severity, causality, and outcome of all SAEs
Dose modifications | Day 1-5
  Dose modifications (incl. reductions and changes in infusion rate)
Time to recovery | Day 29
  Number of days to change to score ≤2 (hospital discharged or meets discharge criteria)
Change over time in ECG parameters | Until day 29
  ECG recordings, (including heart rate, PR interval, RR interval, QRS interval, QT-interval, QTcF) showing abnormal, clinically relevant findings will be reported as adverse event.
Change over time in vital signs | Until day 29
  Changes in recordings of vital sign parameters (including systolic and diastolic blood pressure, Arterial oxygen saturation, heart rate, respiratory rate and body temperature) showing clinically significant measurements outside the normal range will be reported as adverse event.

OTHER OUTCOMES:
Pharmacokinetic assessment of immunoglobulins | Day 1(baseline) to day 29
  Assessment of changes in serum concentrations (g/L) of IgM, IgA, and IgG before, during and after treatment.
Pharmacodynamic assessment of disease related serum proteins | Day 1(baseline) to day 29
  Assessment of relative changes in serum concentrations from baseline before, during and after treatment including inflammation markers (e.g. % change in CRP, PCT, Ferritin, TNF-alpha, IL-6, IL-8 and IL-10), biomarkers (e.g. % change in p-selectin) and complement factors (e.g. % change in C3, C4).

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Torres, MD, Principal Investigator — University of Barcelona Hospital Clinic of Barcelona Spain
Locations (17):
- Brazil (4):
  - Investigational site # 5503, Porto Alegre
  - Investigational site # 5502, Santo André
  - Investigational site # 5505, Santo André
  - Investigational site # 5501, São Paulo
- France (3):
  - Investigational site # 3304, Paris
  - Investigational Site # 3301, Paris
  - Investigational site # 3305, Saint-Etienne
- Russia (8):
  - Investigational site # 0707, Kemerovo
  - Investigational site # 0709, Krasnoyarsk
  - Investigational site # 0702, Moscow
  - Investigational site # 0706, Moscow
  - Investigational site # 0711, Moscow
  - Investigational Site # 0704, Moscow
  - Investigational site # 0708, Moscow
  - Investigational site # 0701, Saint Petersburg
- Spain (2):
  - Investigational Site # 3401, Barcelona
  - Investigational Site # 3402, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Agafina A, Aguiar VC, Rossovskaya M, Fartoukh MS, Hajjar LA, Thiery G, Timsit JF, Gordeev I, Protsenko D, Carbone J, Pellegrini R, Stadnik CMB, Avdeev S, Ferrer M, Heinz CC, Hader T, Langohr P, Bobenhausen I, Schuttrumpf J, Staus A, Ruehle M, Weissmuller S, Wartenburg-Demand A, Torres A. Efficacy and safety of trimodulin in patients with severe COVID-19: results from a randomised, placebo-controlled, double-blind, multicentre, phase II trial (ESsCOVID). Eur J Med Res. 2024 Aug 13;29(1):418. doi: 10.1186/s40001-024-02008-x. PMID 39138518